CLINICAL TRIAL: NCT00494572
Title: Pharmacokinetics and Pharmacodynamics of Montelukast in Children, Ages 6 Through 18 Years Old, With Status Asthmaticus Unresponsive to Conventional Treatment
Brief Title: Montelukast With Status Asthmaticus, Ages 6-18
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Pediatric Pharmacology Research Units Network (Network)
Responsible Party: Jeffrey L. Blumer, Ph.D., M.D., University Hospitals Case Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPRU 10856
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-11

CONDITIONS: Status Asthmaticus; Asthma
Keywords: Montelukast; Albuterol; Status Asthmaticus; Asthma
MeSH Terms: conditions — Status Asthmaticus; Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sterile Water (Sham Comparator): Sterile water
  Interventions: Other: sterile water
- Montelukast (Active Comparator): 10mg rapid dissolving granules in sterile water orally once
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — 10 mg rapid dissolving granule in sterile water orally once
  Arms: Montelukast
Other: sterile water — sterile water
  Arms: Sterile Water

SUMMARY:
The purpose of this study is to determine if montelukast, in addition to standard treatment is helpful in treating patients ages 6-18 who are in the hospital because of status asthmaticus.

DETAILED DESCRIPTION:
This is a prospective study of montelukast efficacy in addition to standard treatment of status asthmaticus in children who are in the PICU. The study will be stratified in 2 groups: children 6-12 years of age and adolescents 13-18 years of age. Children who meet eligibility requirements will be randomized to receive a rapid-dissolving oral dose of montelukast or placebo. Participants will be given a physical exam, have FEV1 measurements and clinical asthma scores recorded pre- and post- completion of a nebulized albuterol treatment of 0.1 mg/kg/dose (min 2.5 mg/dose). Blood samples for PK analysis will be collected prior to study drug administration and at predetermined time intervals to determine the plasma level of montelukast. In addition, a blood sample will be obtained for genetic study of polymorphisms of CYP3A4, CYP3A5, and CYP2C9.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent/legal guardian must give written informed consent and written assent must be obtained form the subject prior to study participation.

  1. Obtain consent of the parent/legal guardian using a signed consent form;
  2. Obtain assent form minors between the ages of 7-13 using a signed assent form;
  3. Obtain assent from minors between the ages of 14-17 by having the subject sign the consent formed signed the parent / legal guardian (Or based on the assessment by the Primary Investigator that the patient is unable to comprehend the study as written in the consent form document, the patient may document assent by signing the assent form).
* Participant, male or female, must be 6 to 18 years of age.
* Participant must have a history of reactive airway disease (RAD) or asthma and must currently be admitted for an acute exacerbation of RAD or asthma.
* Primary physician must believe that patient would benefit from improved bronchodilation and improvement in clinical asthma severity score.
* Participant must have received standard therapy for status asthmaticus:

  1. Oxygen as needed
  2. >3 nebulized albuterol treatments of at least 2.5mg/dose
  3. Methylprednisolone or prednisone loading dose of 2mg/kg
  4. Ongoing methylprednisolone therapy @ 0.5mg/kg every 6 hours
* Participant must have received steroids at least 6 hours prior to their inclusion, and must still require nebulized albuterol at least every 2 hours, as determined by PICU team in accordance with the PICU standard for evaluating and treating patients with RAD or asthma exacerbations.
* Participant must have an indwelling catheter in place from which to obtain blood specimens. Catheter may be peripheral or central, arterial or venous.

Exclusion Criteria:

* Known hypersensitivity to montelukast
* Chronic lung disease other than RAD or asthma
* Known renal disease
* Known hepatic disease
* Cardiac or pulmonary congenital anomalies
* Known immunologic disorders other than allergy and atopy
* Other explanations for respiratory distress
* Use of leukotriene modifiers within 2 weeks of the acute presentation
* Pregnant females
* Intubated patients
* Inability to participate in portable spirometry for FEV1 measurement

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-01 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate effectiveness of Montelukast as adjunctive therapy

SECONDARY OUTCOMES:
Estimate the first dose pharmacokinetic parameter of Montelukast

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Blumer, MD, Principal Investigator — PPRU
Locations (1):
- Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States